CLINICAL TRIAL: NCT05062109
Title: Multimodal Geriatric Pre-authorization Before Scheduled Orthopedic Surgery
Acronym: PRE4OS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-A03323-36
Record Dates: First submitted 2021-08-07; First posted 2021-09-30 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Osteoarthritis; Gonarthrosis
Keywords: osteoarthritis; gonarthrosis; orthopaedic surgery
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multimodal geriatric prehabilitation (Experimental)
  Interventions: Behavioral: Multimodal geriatric prehabilitation

INTERVENTIONS:
Behavioral: Multimodal geriatric prehabilitation — Multimodal prehabilitation will be carried out over a period of 6 weeks in a day admission (once a week) and at home, and will include:
  * Muscle rehabilitation developed with a physiotherapist or physical activity monitor
  * Nutritional support (dietitian at the 1st, 3rd, and 6th day admission (DA))
  * Cognitive and physical stimulation "Exergame"
  * Psychological support by a psychologist
  * Information in the form of videos on the main risks and important points to know and prepare before and after surgery
  * Assessment of patient satisfaction, any limitations encountered, the possible performance of exercises at home and the occurrence of any adverse effects.
  * One session of adapted physical activity at home of one hour per week by a physical trainer from the Siel Bleu association

SUMMARY:
The main objective of this multicentric, prospective and interventional study is to assess the feasibility of multimodal prehabilitation in patients aged 75 years or older with surgical indication for coxarthrosis or severe gonarthrosis

DETAILED DESCRIPTION:
This study consists of a pre-established surgical preparation program in cooperation with physiotherapists or physical activity instructors, dieticians, psychologists, physical therapists and nurses.

This innovative program improves muscle strength, balance and walking of the study patients. It also allows for faster and better recovery of their physical fitness and intellectual abilities after surgery.

These interventions will be performed in day admission (DA) and at home and will consist of training, a diet program to strengthen the muscles and balance of the patients participating in the study.

Patients who agree to participate in the study will receive interventions for 6 weeks prior to surgery, partly in a day hospital and partly at home, including:

* Muscle rehabilitation developed with a physiotherapist or physical activity instructor
* Nutritional support (dietician at 1st, 3rd, and 6th day admission (DA), referring geriatrician)
* Cognitive and physical stimulation "Exergame" (Genious Healthcare); with only cognitive exercises at home
* Psychological support by a psychologist
* Information in the form of videos on the main risks and important points to know and prepare before and after surgery
* 1 follow-up call per week made by the PRE4OS referent between each day admission (DA) to assess patient satisfaction, any limitations encountered, possible exercises at home, the occurrence of possible adverse effects
* 1 hour per week home adapted physical activity session by the Siel Bleu association

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years
* Surgical indication for total hip or knee replacement for hip or knee osteoarthritis.
* Minimum time of 6 weeks between inclusion visit and date of surgery
* Physical (excluding coxarthrosis or knee osteoarthritis) and cognitive capacities to follow a prehabilitation program (assessment by the geriatrician)
* Proximity between place of life and hospital to go to the center for pre-rehabilitation
* Good understanding of the French language
* Benefiting from social coverage
* Have read the information notice and have consented to participate in the study by signing a written consent

Exclusion Criteria:

* Urgent surgery (trauma, acute dislocation)
* Neurocognitive disorders at a moderate or severe stage (Mini Mental State Examination (M.M.S.E) ≤20), or not evaluable and not allowing to participate in the prehabilitation program
* Lack of social coverage (beneficiary or beneficiary)
* Adult persons subject to a legal protection measure (curatorship, guardianship and safeguard of justice)
* Refusal to participate
* Hospitalized patients ( the living space can be the home or thelon term care).

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
80% participation in the number of sessions by at least 80% of the patients included in the study | 6 weeks

SECONDARY OUTCOMES:
Assessment of quality of life according EuroQol- 5 Dimension (EQ-5D) questionnaire | 6 weeks
  The answers given to ED-5D permit to find 243 unique health states or can be converted into EQ-5D index an utility scores anchored at 0 for death and 1 for perfect health
Physical and Cognitive Stimulation Using an Exergame | 6 weeks
  Cognitive and physical stimulation "Exergame" (Genious Healthcare); with realization only of cognitive exercises at home without including minimum and maximum values
Nutritional assessment measuring the Body Mass Index (BMI) | 6 weeks
Assessment of the degree of patient dependence according "Index of Independence in Activities of Daily Living" KATZ scale | 6 weeks
  This is a measurement of the subject's ability to perform activities of daily living independently. The Index ranks adequacy of performance in the six functions of bathing, dressing, toileting, transferring, continence, and feeding. A high score (6) indicates full function (patient independent). 2 or less score, indicates severe functional impairment.(patient very dependent)
Assessment of patient's level of dependence through an appreciation of instrumental activities of daily living according Lawton scale | 6 weeks
  Assessment of older people: Self-maintaining and instrumental activities of daily living without including minimum and maximum values
Assessment of depression according MINI Geriatric depression scale (Mini-GDS) | 6 weeks
  the aim of this score is to identify and assess risk factors for depression in elderly patients without including minimum and maximum values.
  If the score is greater than or equal to 1: high probability of depression. If the score is 0: high probability of no depression.
Assessment of functional status according Short Physical Performance Battery (SPPB) | 6 weeks
Assessment of function and pain after total knee replacement surgery using Oxford Knee Score (OKS) | 6 weeks
  The Oxford Knee Score (OKS) measures the degree of knee pain and functional status of the knee on a scale ranging from 0 to 48:
  Score 0 to 19: May indicate severe arthritis of the knee Score 20 to 29: May indicate moderate to severe knee arthritis Score 30 to 39: May indicate mild to moderate knee arthritis Score 40 to 48: May indicate satisfactory joint function
Assessment of function and pain after total hip replacement using Oxford HIP Score (OHS) | 6 weeks
  The Oxford hip Score (OHS) assesses pain (6 items) and function (6 items) of the hip in relation to daily activities on a scale ranging from 0 to 48:
  Score 0 to 19: May indicate severe hip arthritis Score 20 to 29 May indicate moderate to severe hip arthritis Score 30 to 39 May indicate mild to moderate hip arthritis Score 40 to 48 May indicate satisfactory joint function
Detection of mild cognitive impairment using Montreal Cognitive Assessment (MoCA) | 6 weeks
Screening for undernutrition using Mini Nutritional Assessment (MNA) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Boddaert, MD PhD, Study Chair — Geriatric Perioperative Unit, Pitié-Salpêtrière hospital
Locations (1):
- Geriatric Perioperative Unit, Pitié-Salpêtrière hospital, Paris, IIe-de-France, France